CLINICAL TRIAL: NCT04207710
Title: Study to Determine the Safety of Gebauer's Ethyl Chloride and Gebauer's Pain Ease Sprays When Used Following ChloraPrep for Invasive Procedures
Brief Title: Safety of Gebauer's Pain Ease and Gebauer's Ethyl Chloride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Gebauer Company (Network)
Responsible Party: Principal Investigator, Katherine Nowak, PhD, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12932
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Spray; Pain; Safety Issues
Keywords: Pain Ease; Ethyl Chloride; Safety; Topical anesthetic; ChloraPrep; Topical refrigerant; Microbial growth
MeSH Terms: conditions — Pain | interventions — pain ease refrigerant; Ethyl Chloride

STUDY DESIGN:
Intervention Model Description: 72 participants will have an area of skin on the wrist and lower back swabbed three times each. First, the untreated patch of skin will be swabbed, then it will be treated with ChloraPep and swabbed, then Pain Ease spray will be applied and the area will be swabbed again. The same process will be performed using Ethyl Chloride spray instead of Pain Ease on the opposite wrist and adjacent area on the lower back. The bacterial growth will be compared amongst the different treatments, based on the number of colony forming units that are present.
Who Masked: Outcomes Assessor
Masking Description: The microbiology lab staff culturing and analyzing the samples for microbial growth will not know what type of treatment each sample received. Each sample will only be labelled with a numerical string. The research staff will have a spreadsheet to determine which numerical string corresponds with which treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Microbial growth on wrist after application of Gebauer's Ethyl Chloride (Experimental): An area of skin on the wrist will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Ethyl Chloride topical refrigerant spray. The bacterial growth prior to and after numbing spray application will be evaluated, based on the number of colony forming units that are present.
  Interventions: Drug: Gebauer's Ethyl Chloride
- Microbial growth on lower back after application of Gebauer's Ethyl Chloride (Experimental): An area of skin on the lower back will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Ethyl Chloride topical refrigerant spray. The bacterial growth prior to and after numbing spray application will be evaluated, based on the number of colony forming units that are present.
  Interventions: Drug: Gebauer's Ethyl Chloride
- Microbial growth on wrist after application of Gebauer's Pain Ease (Experimental): An area of skin on the wrist will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Pain Ease topical refrigerant spray. The bacterial growth prior to and after numbing spray application will be evaluated, based on the number of colony forming units that are present.
  Interventions: Drug: Gebauer's Pain Ease Top Aerosol Mist Spray
- Microbial growth on lower back after application of Gebauer's Pain Ease (Experimental): An area of skin on the lower back will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Pain Ease topical refrigerant spray. The bacterial growth prior to and after numbing spray application will be evaluated, based on the number of colony forming units that are present.
  Interventions: Drug: Gebauer's Pain Ease Top Aerosol Mist Spray

INTERVENTIONS:
Drug: Gebauer's Pain Ease Top Aerosol Mist Spray — Topical refrigerant spray
  Other Names: Pain Ease
  Arms: Microbial growth on lower back after application of Gebauer's Pain Ease; Microbial growth on wrist after application of Gebauer's Pain Ease
Drug: Gebauer's Ethyl Chloride — Topical refrigerant spray
  Other Names: Ethyl Chloride
  Arms: Microbial growth on lower back after application of Gebauer's Ethyl Chloride; Microbial growth on wrist after application of Gebauer's Ethyl Chloride

SUMMARY:
This study aims to determine if Gebauer's Pain Ease or Gebauer's Ethyl Chloride topical anesthetic sprays are safe for use as numbing agents prior to placing epidurals and arterial lines, based on whether they introduce increased microbial growth after application to skin. Due to the recent national shortage of lidocaine, we hope to find a suitable alternative to lidocaine for topical analgesia when placing arterial lines and epidurals. Our hypothesis is that the sprays will not affect the sterility of the area. We will compare microbial growth from three subsequent swabs taken from a single area of skin on the wrist and lower back: one with no treatment, the second after treatment with ChloraPrep, and the third after applying one of the numbing sprays. If there is significantly higher growth in the swabs containing the topical anesthetic spray versus the ChloraPrep alone, this will indicate that the sprays introduce microbes to the sites of skin.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether Gebauer's Pain Ease and Ethyl Chloride topical anesthetic sprays are safe for application on the areas of skin where epidurals (lower back) and arterial lines (wrist) are placed, based on whether they introduce microbial growth to these areas. The investigators will compare microbial growth by swabbing both of these skin sites following: 1) no treatment 2) ChloraPrep treatment and 3) ChloraPrep plus numbing spray (Ethyl Chloride or Pain Ease) treatment. The cultures will then be incubated to test for anaerobic bacteria, aerobic bacteria, and mold growth. The microbial growth will be compared between the three treatment groups based on the number of colony forming units present.

Funding for the project will be from the manufacturer of the numbing sprays, Gebauer Company.

Based on power analysis, for each of the numbing sprays, a total of 72 subjects must be enrolled, with 6 swabs taken per subject (untreated, ChloraPrep, and topical anesthetic spray samples will be taken from both the wrist and lower back of each subject). A sample size of 72 pairs achieves 80 % power to detect an odds ratio of 24 using a two-sided McNemar test with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Henry Ford employees

Exclusion Criteria:

* People with infections at the site of prep
* People with history of hypersensitivity to numbing sprays or chloraprep

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mlynek K, Lyahn H, Richards B, Schleicher W, Bassiri Gharb B, Procop G, Tuohy M, Zins J. Skin Sterility After Application of a Vapocoolant Spray Part 2. Aesthetic Plast Surg. 2015 Aug;39(4):597-601. doi: 10.1007/s00266-015-0509-5. Epub 2015 Jun 5. PMID 26044395
- [Background] Polishchuk D, Gehrmann R, Tan V. Skin sterility after application of ethyl chloride spray. J Bone Joint Surg Am. 2012 Jan 18;94(2):118-20. doi: 10.2106/JBJS.K.00229. PMID 22257997

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: patch of skin
Groups:
- Microbial Growth on Wrists and Lower After Application of Gebauer's Ethyl Chloride or Pain Ease.: An area of skin on the wrist swabbed before and after Chloraprep application, and then each area swabbed again after application of Gebauer's Ethyl Chloride topical refrigerant spray. Bacterial growth prior to and after numbing spray application evaluated, based on number of colony forming units present.
  An area of skin on the lower back of an individual's skin swabbed before and after Chloraprep application, and then each area swabbed again after application of Gebauer's Ethyl Chloride topical refrigerant spray. Bacterial growth prior to and after spray application evaluated, based on number of colony forming units present.
  An area of skin on the wrist swabbed before and after Chloraprep application, and then swabbed again after application of Gebauer's Pain Ease topical refrigerant spray. Bacterial growth prior to and after spray application evaluated, based on number of colony forming units present.
  An area of skin on the lower back swabbed before and after Chloraprep application, and then after application of Gebauer's Pain Ease topical refrigerant spray. Bacterial growth prior to and after spray application evaluated, based on number of colony forming units present.
Period: Overall Study
Arm/Group | Microbial Growth on Wrists and Lower After Application of Gebauer's Ethyl Chloride or Pain Ease.
Started | 72; 288 patch of skin
Left Wrist: ChloraPrep, Then Gebauer's Ethyl Chloride | 72; 72 patch of skin
Right Wrist: ChloraPrep, Then Gebauer's Pain Ease | 72; 72 patch of skin
Low Back: ChloraPrep, Then Gebauer's Ethyl Chloride | 72; 72 patch of skin
Low Back: ChloraPrep, Then Gebauer's Pain Ease | 72; 72 patch of skin
Completed | 72; 288 patch of skin
Not Completed | 0; 0 patch of skin

BASELINE CHARACTERISTICS:
Groups:
- Microbial Growth on Skin After Application of Gebauer's Ethyl Chloride or Pain Ease: In a split-person design, each subject had four areas of skin swabbed as follows:
  * Left wrist swabbed before and after Chloraprep application, and again after application of Gebauer's Ethyl Chloride topical refrigerant spray
  * Right wrist swabbed before and after Chloraprep application, and again after application of Gebauer's Pain Ease.
  * Low back swabbed before and after Chloraprep application, and then after application of Gebauer's Ethyl Chloride topical refrigerant spray.
  * Another section of low back swabbed before and after Chloraprep application, and then after application of Gebauer's Pain Ease topical refrigerant spray.
  The bacterial growth prior to and after numbing spray application were evaluated based on the number of colony forming units that were present.
Arm/Group | Microbial Growth on Skin After Application of Gebauer's Ethyl Chloride or Pain Ease
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age information was not collected as this was irrelevant to the study aims.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender information was not collected for this study as it was not relevant to the study aims.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Presence of Microbial Growth (1+ CFU)
Description: Number of skin samples that were positive for bacterial growth following treatment with ChloraPrep and then application of a topical refrigerant spray (Gebauer's Ethyl Chloride or Gebauer's Pain Ease), when the area was swabbed and cultured for three days. A sample was considered positive if 1 or more colony forming units were present per swab.
Time Frame: Skin samples were swabbed within 20 seconds of Ethyl Chloride or Pain Ease application, and then swabs were cultured for 3 days before checking for the presence of CFU.
Measure: Number; unit: Number of samples with 1+ CFU
Groups:
- Wrist, Gebauer's Ethyl Chloride: Skin on wrist swabbed before treatment, then following sterilization with Chloraprep, then after treatment with Gebauer's Ethyl Chloride topical refrigerant spray. Samples cultured and evaluated for positive bacterial growth.
- Lower Back, Gebauer's Ethyl Chloride: Skin on lower back swabbed before treatment, then after sterilization with Chloraprep, then after application of Gebauer's Ethyl Chloride topical refrigerant spray. Samples cultured and evaluated for positive bacterial growth.
- Wrist, Gebauer's Pain Ease: Wrist swabbed before treatment, after sterilization with Chloraprep, then after application of Gebauer's Pain Ease. Samples cultured and evaluated for positive bacterial growth.
- Lower Back, Gebauer's Pain Ease: Lower back swabbed before treatment, after Chloraprep, then after application of Gebauer's Pain Ease. Samples cultured and evaluated for positive bacterial growth.
Arm/Group | Wrist, Gebauer's Ethyl Chloride | Lower Back, Gebauer's Ethyl Chloride | Wrist, Gebauer's Pain Ease | Lower Back, Gebauer's Pain Ease
Number analyzed (Participants) | 72 | 72 | 72 | 72
Number of samples with 1+ CFU
  Samples with positive growth after application of ChloraPrep followed by topical refrigerant spray | 2 | 1 | 1 | 1
  Samples with positive growth after application of ChloraPrep | 1 | 0 | 0 | 2
  Samples with positive growth before ChloraPrep treatment (positive control) | 68 | 63 | 65 | 49
Statistical Analysis 1: Comparison: Wrist, Gebauer's Ethyl Chloride; Comparison of incidence of positive growth in samples obtained following application of ChloraPrep vs. ChloraPrep followed by Gebauer's Ethyl Chloride; Test type: Superiority; p = 0.317, Friedman — A priori threshold for significance was p<0.05
Statistical Analysis 2: Comparison: Lower Back, Gebauer's Ethyl Chloride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.317, Friedman — A priori threshold was p<0.05
Statistical Analysis 3: Comparison: Wrist, Gebauer's Pain Ease; Comparison of incidence of positive growth in samples obtained following application of ChloraPrep vs. ChloraPrep followed by Gebauer's Pain Ease; Test type: Superiority; p = 0.317, Friedman — A priori threshold was p<0.05
Statistical Analysis 4: Comparison: Lower Back, Gebauer's Pain Ease; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.317, Friedman — A priori threshold was p<0.05

ADVERSE EVENTS:
Time Frame: During swabbing of skin (5-15 minutes)
Groups:
- Microbial Growth on Lower Back After Application of Gebauer's Ethyl Chloride: An area of skin on the lower back of an individual's skin will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Ethyl Chloride topical refrigerant spray. The bacterial growth prior to and after spray application will be evaluated, based on the number of colony forming units that are present.
- Microbial Growth on Wrist After Application of Gebauer's Pain Ease: An area of skin on the wrist of an individual's skin will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Pain Ease topical refrigerant spray. The bacterial growth prior to and after spray application will be evaluated, based on the number of colony forming units that are present.
- Microbial Growth on Lower Back After Application of Gebauer's Pain Ease: An area of skin on the lower back of an individual's skin will be swabbed before and after Chloraprep application, and then each area will be swabbed again after application of Gebauer's Pain Ease topical refrigerant spray. The bacterial growth prior to and after spray application will be evaluated, based on the number of colony forming units that are present.
Arm/Group | Microbial Growth on Wrist After Application of Gebauer's Ethyl Chloride | Microbial Growth on Lower Back After Application of Gebauer's Ethyl Chloride | Microbial Growth on Wrist After Application of Gebauer's Pain Ease | Microbial Growth on Lower Back After Application of Gebauer's Pain Ease
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04207710/Prot_SAP_000.pdf